CLINICAL TRIAL: NCT06063928
Title: Confronting Cancer as a Community
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3C-21-3; NCI-2022-10775 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 3C-21-3 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH); U2CCA252971 (NIH)
Record Dates: First submitted 2023-09-06; First posted 2023-10-03 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Usual Care (Experimental): Patients will receive standard educational materials prior to the return of their results to better understand the results.
  Interventions: Other: Usual Care Educational Materials
- Arm 2: Intervention (Experimental): Patients will receive CoGenes educational materials and video prior to the return of their results to better understand the results. The goal is to provide education about the benefits of genetic and tumor testing and to increase the patient's knowledge.
  Interventions: Other: Intervention Educational Materials

INTERVENTIONS:
Other: Usual Care Educational Materials — Standard education materials
  Arms: Arm 1: Usual Care
Other: Intervention Educational Materials — CoGenes educational materials with video.
  Arms: Arm 2: Intervention

SUMMARY:
This study aims to better understand the cause of colorectal cancer and how to find the best treatment for Hispanic patients with colorectal cancer. The genetic information in the blood and tissues may explain why patients who have the same type of cancer and receive the same treatment do not always have the same results. By combining genetic (certain qualities or traits passed from parents to offspring) information with clinical data, such as the responses of different kinds of cancers to different treatments, this study could lead to more knowledge about why certain cancers occur and why they respond differently to treatments. Information gathered from this study may help researchers match treatments to the genetics of each patient and the genetic changes in their tumor. This approach is known as personalized medicine.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To create a well-characterized cohort of Hispanic patients with colon cancer, with patient-level data, genomic, transcriptomic, clinical, and outcomes data.

SECONDARY OBJECTIVES:

I. To identify genomic/transcriptomic predictors of treatment outcomes (time to recurrence, time to progression, and overall survival).

II. To identify associations between somatic tumor deoxyribonucleic acid (DNA) methylation patterns and clinical outcomes.

III. To examine patterns of patient engagement in genetic/genomic testing among Hispanic patients with colorectal cancer (CRC).

IV. To compare two strategies for providing education to patients before receiving genetic results.

EXPLORATORY OBJECTIVES:

I. To validate, characterize and discover molecular processes in the CRC tumor common to other CRC populations and specific to Hispanic patients.

II. To determine whether comorbidities are associated with variation in tumor molecular pathways and whether comorbidities are effect modifiers of associations between tumor molecular variation and disease outcomes and response to treatment in Hispanic CRC patients.

III. To perform microbiome sequencing through a stool collection kit and nucleic acid extraction to understand the interplay between gut microbiome and cancer progression and response to therapy.

IV. Conduct in-depth analysis of the gut microbiome in the context of genomic characterization and clinical variables.

V. Evaluate the impact of conducting genetic and tumor testing among colorectal cancer patients in the clinic.

VI. Evaluate associations between lifestyle, dietary, and social determinants of health and clinical outcomes and tumor characteristics.

VII. Identify potential reasons why some participants decline to participate in this study.

VIII. Increase understanding of family communication of germline test results.

IX. Explore the barriers to and facilitators of cascade testing among participants who have a germline pathogenic variant.

OUTLINE: This is an interventional study.

Patients undergo blood sample collection, collection of archival tumor tissue and genetic testing, and complete questionnaires on study. Patients also have their medical records reviewed on study. Patients are randomized into one of two arms before they receive their test results -- Arm 1: Usual Care and Arm 2: Intervention.

After return of genetic testing results, patients are followed up at 2 weeks, 6 months (one blood draw), 12 months, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Hispanic ethnicity
* Diagnosed with colon or rectal cancer (at any time and stage; lifetime diagnosis and in survival are eligible)
* Has a tumor tissue sample archived or plans to have tissue archived from a standard care procedure
* Age >= 18 years
* Ability to understand and the willingness to sign a written informed consent.
* For those who would like to participate in the optional microbiome characterization aspect of the study, the patient will have to be under 40 years old at any clinical cancer stage or over 60 years old at any clinical cancer stage.

Exclusion Criteria:

* Inability to understand and the willingness to sign a written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2027-05-25 (Estimated); Study Completion 2028-05-25 (Estimated)

PRIMARY OUTCOMES:
Time to recurrence (TTR) | Assessed up to 6 years
  Determined from time of registration to date of documented event such as treatment-related deaths, second same or other primary cancers, and deaths from other cancers.
Progression free survival (PFS) | Assessed up to 6 years
  Determined from start of treatment to time of progression or death (whichever comes first).
Overall survival (OS) | Assessed up to 6 years
  Determined from start of treatment until death due to any cause.
Changes in genomic knowledge | Baseline, at 2 weeks, and at 12-month follow up
  The KnowGene scale will be used. Score Range = 0-16. Higher score indicates higher knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Lenz, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California